CLINICAL TRIAL: NCT00493545
Title: A Multicenter, Nonrandomized, Open-Label Phase 1 Safety Study of HspE7 and Poly-ICLC Administered Concomitantly in Cervical Intraepithelial Neoplasia (CIN) Subjects
Brief Title: Safety Study to Test the Safety of HspE7 and Poly-ICLC Given in Patients With Cervical Intraepithelial Neoplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nventa Biopharmaceuticals Corporation (Industry)
Responsible Party: Dr. Peter Emtage Vice President of Research and Development, Nventa Biopharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HspE7-00101-0601
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Multicenter; Open-Label; Nonrandomized; Safety
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: HspE7 and Poly-ICLC — 3 injections of HspE7 and Poly ICLC given every 28 days for 3 injections

SUMMARY:
The purpose of this study is to determine the safety and tolerability of HspE7 and Poly-ICLC when given together

DETAILED DESCRIPTION:
Approximately 600 million people worldwide are infected with the Human Papilloma Virus. In the majority of cases people can clear the virus on their own however in cases where the infection is not recognized or is left untreated, the result can be cervical cancer.

This study will examine the safety and tolerability of Hsp-E7 and Poly-ICLC administered together as a vaccine for Cervical Intraepithelial neoplasia (CIN). There will be 4 cohorts of subjects in the study each given a higher dose than the one prior providing that prior dose has been well tolerated and deemed to be safe.

Subjects will be immunized every 28 days for a period of 8 weeks (3 administrations).

Posttreatment evaluation will occur 4 weeks after the last of 3 injections. Subjects with CIN 2 or 3 disease at the time of enrollment will be eligible to undergo clinically appropriate therapeutic treatment of the cervix at the twelfth of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented Cervical Intraepithelial Neoplasia 1, 2 or 3.
2. Nonpregnant, Nonlactating female greater than or equal to 18 years of age, who is either surgically sterile, postmenopausal (no menses for the previous 12 months), or practices an effective method of birth control (to be continued throughout the study period) as determined by the Investigator (eg: oral contraceptives, injectables or implants, intrauterine device, double-barrier methods). The use of cervical cap or diaphram is not permitted).
3. Geographically accessible for ongoing follow up and committed to comply with all visits.
4. Judged to be in good health based upon the results of a medical history, physical examination, vital signs and laboratory profile.
5. Capable of understanding and complying with the protocol and has signed the informed consent.
6. Negative for human immunodeficiency virus (HIV)-1, HIV-2, Hepatitis B surface antigen, and hepatitis C Virus.

Exclusion Criteria:

Prior to Therapy:

1. Prior exposure to HspE7.
2. The subject received immunotherapy (eg, interferons, tumor necrosis factor, interleukins, or biological response modifiers [GM CSF, G CSF, M CSF]) within 4 weeks (28 days) prior to study entry.
3. Taken within 7 days or is currently taking selective Cox-2 inhibitors and other nonsteroidal anti-inflammatory drugs.
4. Received investigational systemic drugs within 4 weeks (28 days) prior to study entry.
5. Undergoing active treatment of genital warts.
6. Has taken astemizole within 7 days prior to study drug administration.

Disease Status:

1. Has an autoimmune disease that in the opinion of the investigator would compromise the safety of the subject in this study. Some examples of autoimmune disease that may be considered exclusionary include rheumatoid arthritis, systematic lupus erythematosus, and autoimmune thyroiditis.
2. Has a recognized immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia. The subject has hereditary or congenital immunodeficiencies.
3. Has a positive endocervical curettage at the time of biopsy.

Physiological Functions:

1. Has clinically significant hepatic dysfunction (ie, alanine aminotransferase, aspartate aminotransferase, or total bilirubin ≥1.5 x upper limit of normal (ULN).
2. Has clinically significant renal dysfunction (ie, serum creatinine ≥1.5 x ULN).
3. Has clinically significant cardiac disease, eg, New York Heart Association classes III IV, uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, or myocardial infarction in the previous 6 months as confirmed by an electrocardiogram.
4. Has had a splenectomy.
5. Has an infectious process that in the opinion of the investigator would compromise the subject's ability to mount an immune response.
6. Has a history of severe allergic reaction to insect bites or stings, or to any biologic pharmaceutical product, including compounds similar to the test article.
7. Has donated or lost a significant volume of blood or plasma (greater than 450 mL) within 30 days of the study.

Standard Safety:

1. Is pregnant or breast-feeding, or a woman of childbearing potential unless using effective contraception as determined by the investigator. Subjects whom the investigator considers may be at risk of pregnancy will have a pregnancy test performed per institutional standard.
2. Any other reason that, in the opinion of the investigator, precludes the subject from participating in the study.
3. Known hypersensitivity reaction to any of the components of study treatments.
4. Known alcohol or drug abuse, as assessed by the investigator.
5. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Safety of HspE7 and Poly-ICLC administered concomitantly for Cervical Intraepithelial Neoplasia | 4 Weeks after the last of 3 Injections

SECONDARY OUTCOMES:
Tolerability of HspE7 and Poly-ICLC administered concomitantly for Cervical Intraepithelial Neoplasia | 4 Weeks after the last of 3 Injections

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Medical Center for Clinical Research, San Diego, California
  - Medical College of Georgia, Augusta, Georgia
  - Montefiore Medical Center, New York, New York
  - University of Oklahoma Health Sciences Center (OUHSC) / OU Medical Center, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - Mt Timpanagos Women's Health Center, Pleasant Grove, Utah
  - Salt Lake Women's Center, South Salt Lake, Utah